CLINICAL TRIAL: NCT03691298
Title: Prospective, Multicenter, Post-Market 1 Year Clinical Follow-up Study to Evaluate Safety and Performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in Shoulder and Hip Arthroscopic Repair
Brief Title: Safety and Performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in Shoulder and Hip Arthroscopic Repair
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: 17-5010-06
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2022-06

CONDITIONS: Instability, Joint
Keywords: Suturefix; hip instability; shoulder instability
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic hip and shoulder repair
  Interventions: Device: SUTUREFIX ULTRA Suture Anchor and SUTUREFIX CURVED Suture Anchor

INTERVENTIONS:
Device: SUTUREFIX ULTRA Suture Anchor and SUTUREFIX CURVED Suture Anchor — Fixation device intended to provide secure fixation of soft tissue to bone

SUMMARY:
The scientific justification is to fulfill post-market clinical requirements in order to support re-certification of the CE-Mark for this marketed product and to look into safety and efficacy.

DETAILED DESCRIPTION:
Shoulder: The superior labrum (fibrous cartilage) and biceps anchor improve joint stability by acting like a secondary stabilizer to the shoulder. Labral injuries are usually associated with anterior shoulder dislocation. When conservative treatment fails, such as physical therapy, strengthening programs, anti-inflammatories and activity modification to improve symptoms, surgical intervention may be required. Surgical treatments can include simple debridement, stabilization of the biceps-labrum complex through repair, or biceps tenodesis where the end of a tendon is joined surgically to the bone. Outcomes of SLAP (superior labral tear from anterior to posterior) repairs have been reported good throughout the literature, with reported success rates ranging from 71-97%.

Hip: The labrum of the hip is a fibrocartilaginous tissue that connects to the bone edge of the acetabulum (the socket of the hip bone), and deepens the acetabular socket while extending coverage of the femoral head; it also aids in hip stabilization. The goal of surgical intervention is to restore normal hip mechanics and treat existing damage.

ELIGIBILITY:
Inclusion Criteria:

* Subject has consented to participate in the study by signing the EC-approved informed consent form
* Subject condition meets proposed indication to SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchor
* Subject requiring shoulder or hip arthroscopic labral repair surgery from physical findings, subject symptoms and radiographic finding
* Hip subjects only:

  * FAI (Femoroacetabular Impingement)
* Shoulder subjects only:

  * Subject with a history of recurrent dislocation/subluxation of the shoulder

Exclusion Criteria:

* Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1 (pre-operative)
* Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures
* Contraindications or hypersensitivity to the use of the SUTUREFIX ULTRA and/or SUTUREFIX CURVED Suture Anchor, or their components (e.g. silicone, polyester). Where material sensitivity is suspected, appropriate tests should be performed and sensitivity ruled out prior to implantation
* Pathological conditions of bone, such as cystic changes or severe osteopenia, which would compromise secure anchor fixation
* Pathological conditions in the soft tissues to be attached that would impair secure fixation by suture
* Comminuted bone surface, which would compromise secure anchor fixation
* Hip subjects only:

  * Dysplasia latera/central less than 20°
* Shoulder subjects only:

  * Glenoid and/or humeral bone loss considered excessive by the treating orthopaedic surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with hip or shoulder instability
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Everson, Study Chair — Smith & Nephew Ltd
Locations (9):
- United States (2):
  - New York University Langone Orthopaedic Center, New York, New York
  - Orthotennessee, Knoxville, Tennessee
- CPH Privathospital, Farum, Denmark
- Pihlajalinna Turku Hospital, Turku, Finland
- Azienda Ospedaliera San Camillo Forlanini, Roma, Italy
- Spain (2):
  - Asepeyo Hospital Sant Cugat, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
- United Kingdom (2):
  - Queen Alexandra Hospital, Cosham
  - Fortius Clinic, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled form 07 November 2018 to 21 May 2021.
Pre-assignment Details: Overall, 83 participants (42 hips / 41 shoulders) were enrolled and received the investigational product (IP) at 9 sites.
Period: Overall Study
Arm/Group | Arthroscopic Hip and Shoulder Repair
Started | 83
Completed | 73
Not Completed | 10
Not completed — Lost to Follow-up | 8
Not completed — Sponsor terminated study | 2

BASELINE CHARACTERISTICS:
Population: Data available from the Safety Population (SAF) included all participants that received the investigational product (IP).
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.70 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Black | 2
  Race: Other | 2
  Race: White | 78
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.40 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success at 6 Months
Description: Number of participants without signs of failure and/or re-intervention as assessed by the surgeon.
Time Frame: 6 month post-surgery
Population: Participants from the Full Analysis Set (FAS) utilized for this assessment. Population included participants with available data that were enrolled into the study and attended at least one post-Baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 58
Participants | 56

2. Secondary Outcome: Clinical Success at 12 Months
Description: Number of participants without signs of failure and/or re-intervention at 12 months, as assessed by the surgeon.
Time Frame: 12 months post-operative
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 67
Participants | 64

3. Secondary Outcome: Intra-operative Anchor Deployment Success
Description: Number of suture anchors that were successfully deployed to bone, soft tissues, or both.
Time Frame: Intraoperatively
Population: as for outcome 1
Measure: Count of Units; unit: suture anchors
Units Other Than Participants: suture anchors
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 83
Number analyzed (suture anchors) | 84
suture anchors | 73

4. Secondary Outcome: Intraoperative Suture Anchor Failure
Description: Suture anchor failures categorized by number of participants with:
  * Intra-operative failures (Yes/No)
  * Anchors pulled out (Yes/No)
  * Additional anchors used as a result of failure (Yes/No)
Time Frame: Intraoperatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 73
Participants
  Participants with intra-operative failures: Yes | 6
  Participants with intra-operative failures: No | 67
  Participants with anchors pulled out: number analyzed (Participants) | 29
  Participants with anchors pulled out: Yes | 4
  Participants with anchors pulled out: No | 25
  Participants with additional anchors used as a result of failure: number analyzed (Participants) | 28
  Participants with additional anchors used as a result of failure: Yes | 5
  Participants with additional anchors used as a result of failure: No | 23

5. Secondary Outcome: Device-related Re-Intervention
Description: Number of participants with a device-related adverse event (AE) that required a re-intervention due to the device-related AE.
Time Frame: 12 months
Population: Participants from the Safety Population (SAF) utilized for this assessment. SAF included participants that received the investigational product (IP). Additionally, this assessment only included participants from the SAF population with a device-related adverse event (AE).
Measure: Count of Participants; unit: Participants
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 5
Participants | 1

6. Secondary Outcome: Visual Analog Scale (VAS) Pain Score - All Participants
Description: Assessed participant pain using Visual Analog Scale (VAS) assessments taken 6 and 12 months postoperative intervals. The VAS Pain Score was based on a scale of 0 to 10, with 0 representing no pain and 10 the worst possible pain.
  Note: This Patient Reported Outcome (PRO) was optional and used according to the surgeon's preference.
Time Frame: 6 and 12 months postoperative
Population: Participants from the Full Analysis Set (FAS) utilized for this assessment. Population included participants with available data that were enrolled into the study and attended at least one post-Baseline assessment for the time frames specified.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 58
score on a scale
  6 Months Postoperative | 2.0 (2.38)
  12 Months Postoperative: number analyzed (Participants) | 42
  12 Months Postoperative | 1.0 (1.80)

7. Secondary Outcome: Visual Analog Scale (VAS) Satisfaction Score - All Participants
Description: Assessed participant satisfaction using a Visual Analog Scale (VAS) assessments taken at 6 and 12 month postoperative intervals. The VAS Subject Satisfaction Questionnaire was based on a scale of 0 to 10, with 0 representing very satisfied and 10 very unsatisfied.
  This Patient Reported Outcome (PRO) was optional and used according to the surgeon's preference.
Time Frame: 6 and 12 months postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 58
score on a scale
  6 Months Postoperative | 2.30 (3.26)
  12 Months Postoperative: number analyzed (Participants) | 42
  12 Months Postoperative | 1.0 (1.81)

8. Secondary Outcome: Analysis of EQ-5D-5L Index - All Participants
Description: The EQ-5D-5L Index Score was based on a scale of 0 to 1, with higher index values indicating better health and lower index values indicating worse health.
  This Patient Reported Outcome (PRO) was optional and used according to the surgeon's preference.
Time Frame: 6 months and 12 months postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Hip and Shoulder Repair
Number analyzed (Participants) | 57
score on a scale
  6 Months Postoperative | 0.8 (0.22)
  12 Months Postoperative: number analyzed (Participants) | 52
  12 Months Postoperative | 0.9 (0.20)

9. Secondary Outcome: Analysis of Hip Outcome Score Activities of Daily Living (HOOS-ADL) - Hip Participants
Description: The Hip Outcome Score Activities of Daily Living (HOOS-ADL) Score included 5 domains (Symptoms, Pain, Daily Living, Sport & Recreation and Quality of Life) each assessed at 6 and 12 months postoperative. Each HOOS domain range was based on a scale of 0 to 100, where 0 represents extreme symptoms and 100 represents no symptoms.
Time Frame: 6 and 12 months postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arthroscopic Hip Repair: SUTUREFIX ULTRA Suture Anchor and SUTUREFIX CURVED Suture Anchor: Fixation device intended to provide secure fixation of soft tissue to bone
Arm/Group | Arthroscopic Hip Repair
Number analyzed (Participants) | 35
score on a scale
  6 Months Postoperative: Symptoms: number analyzed (Participants) | 30
  6 Months Postoperative: Symptoms | 74.5 (23.57)
  6 Months Postoperative: Pain: number analyzed (Participants) | 30
  6 Months Postoperative: Pain | 77.8 (22.87)
  6 Months Postoperative: Daily Living: number analyzed (Participants) | 30
  6 Months Postoperative: Daily Living | 85.1 (20.72)
  6 Months Postoperative: Sports and Recreation: number analyzed (Participants) | 30
  6 Months Postoperative: Sports and Recreation | 71.3 (26.34)
  6 Months Postoperative: Quality of Life: number analyzed (Participants) | 30
  6 Months Postoperative: Quality of Life | 64.2 (28.33)
  12 Months Postoperative: Symptoms | 75.7 (23.08)
  12 Months Postoperative: Pain | 78.6 (20.72)
  12 Months Postoperative: Daily Living | 84.0 (21.10)
  12 Months Postoperative: Sports and Recreation | 72.3 (29.21)
  12 Months Postoperative: Quality of Life | 64.5 (28.79)

10. Secondary Outcome: Modified Harris Hip Score (mHHS) - Hip Participants
Description: The Modified Harris Hip Score (mHHS) is a measurement of dysfunction; the higher the score, the better the outcome. The mHHS score range was as follows:
  * <70 (poor result)
  * 70-79 (fair result)
  * 80-89 (good result)
  * >90 (excellent result)
  This Patient Reported Outcome (PRO) was optional and used according to the surgeon's preference.
Time Frame: Preoperative, 6 and 12 months Postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Hip Repair
Number analyzed (Participants) | 38
score on a scale
  Preoperative | 51.3 (17.13)
  6 Months Postoperative: number analyzed (Participants) | 30
  6 Months Postoperative | 71.2 (19.24)
  12 Months Postoperative: number analyzed (Participants) | 35
  12 Months Postoperative | 71.9 (17.88)

11. Secondary Outcome: Rowe Score - Shoulder Participants
Description: The Rowe Scores address categories of shoulder stability, motion, and function. Scores range from 0 to 100 with a score of 90 to 100 points indicating an excellent evaluation, 75 to 89 points indicating a good evaluation, 51 to 74 points indicating a fair evaluation, and 0 to 50 points indicating a poor evaluation.
  This Patient Reported Outcome (PRO) was optional and used according to the surgeon's preference.
Time Frame: 6 and 12 months postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arthroscopic Shoulder Repair: SUTUREFIX ULTRA Suture Anchor and SUTUREFIX CURVED Suture Anchor: Fixation device intended to provide secure fixation of soft tissue to bone
Arm/Group | Arthroscopic Shoulder Repair
Number analyzed (Participants) | 28
score on a scale
  6 Months Postoperative: number analyzed (Participants) | 23
  6 Months Postoperative | 93.3 (11.54)
  12 Months Postoperative | 97.9 (8.54)

12. Secondary Outcome: American Shoulder and Elbow Surgeons Score - Shoulder Participants
Description: The American Shoulder and Elbow Surgeons Score (ASES) was based on a scale of 0 to 100 points, where 0 indicated a worse shoulder condition and 100 indicated a better shoulder condition
Time Frame: 6 and 12 months postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Shoulder Repair
Number analyzed (Participants) | 32
score on a scale
  6 Months Postoperative: number analyzed (Participants) | 28
  6 Months Postoperative | 91.0 (12.15)
  12 Months Postoperative | 95.7 (7.99)

13. Secondary Outcome: Constant-Murley Shoulder Scores (CMS) - Shoulder Participants
Description: The Constant-Murley Shoulder Score (CMS) was based on a scale of 0 to 100 points divided into 4 subscales; pain (15 points), Activities of Daily Living (20 points), strength (25 points), and Range of Motion, including: forward elevation, external rotation, abduction, and internal rotation (40 points). The higher the score, the higher the quality of the function (less disability).
Time Frame: 6 months and 12 months Postoperative
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arthroscopic Shoulder Repair
Number analyzed (Participants) | 28
score on a scale
  6 Months Postoperative: number analyzed (Participants) | 23
  6 Months Postoperative | 77.9 (5.95)
  12 Months Postoperative | 79.8 (3.63)

ADVERSE EVENTS:
Time Frame: Time of surgery through 12 months postoperative visit
Description: Adverse Events (AEs) and Device Deficiencies (DDs) were reported and assessed by the Investigators and were additionally analysed and classified by the Sponsor. All AEs presented were finalized on the Adverse Event Monitoring Board (AEMB) Sponsor classifications. This independent review was conducted per ISO 14155 standards. Both the Investigator AE assessment and the Smith+Nephew AEMB independent safety review are included.
Arm/Group | Arthroscopic Hip and Shoulder Repair
All-Cause Mortality (participants affected / at risk) | 0/83
Serious Adverse Events (participants affected / at risk) | 4/83
Other Adverse Events (participants affected / at risk) | 13/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arthroscopic Hip and Shoulder Repair (N=83)
POSTRAUMATIC DISLOCATION LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
INCREASED PAIN RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
NERUOPRAXIA AND PAIN (Nervous system disorders) | 1
RECURRENT INSTABILITY (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arthroscopic Hip and Shoulder Repair (N=83)
ACUTE PAIN RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1
HIP HURTING AND CLICKING INTERMITTENTLY (Musculoskeletal and connective tissue disorders) | 1
GUARDING AROUND LEFT HIP ON EXAMINATION (Musculoskeletal and connective tissue disorders) | 1
MISLOCATION OF DEVICE / LABRUM FAILURE (Musculoskeletal and connective tissue disorders) | 1
INCREASED PAIN 7 MONTHS POST OP (Musculoskeletal and connective tissue disorders) | 1
INCREASED PAIN 3 MONTHS POST OP (Musculoskeletal and connective tissue disorders) | 1
NUMBNESS OF OPER FOOT (Nervous system disorders) | 1
TISSUE DAMAGE (Musculoskeletal and connective tissue disorders) | 2
PARTIAL PARONEAL NERVE PARESIS (Nervous system disorders) | 2
RIGHT SHOULDER STIFFNESS. (Musculoskeletal and connective tissue disorders) | 1
GLENOHUMERAL OSTEOARTHRITIS IN RIGHT S. (Musculoskeletal and connective tissue disorders) | 1
CORONA VIRUS / COVID (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
COVID-19 pandemic impacted the study causing delays on obtaining outcome and safety data at follow-up visits for participants due to site closures and/or site restrictions. There was also an impact on participant retention due to the pandemic with participants being lost to follow-up and/or out of window visits leading to protocol deviations. Patient Reported Outcomes (PROs) were optional & used according to surgeon preference leading to low response rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03691298/Prot_SAP_000.pdf